CLINICAL TRIAL: NCT02576275
Title: A Phase 3, Randomized, Double-blind Study of Duvelisib Administered in Combination With Rituximab and Bendamustine vs Placebo Administered in Combination With Rituximab and Bendamustine in Subjects With Previously-Treated Indolent Non-Hodgkin Lymphoma
Brief Title: A Study of Duvelisib in Combination With Rituximab and Bendamustine vs Placebo in Combination With Rituximab and Bendamustine in Subjects With Previously-Treated Indolent Non-Hodgkin Lymphoma (BRAVURA)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The scope of the program has been reduced to focus resources on studies which can potentially enable the registration of duvelisib.
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPI-145-22
Record Dates: First submitted 2015-10-07; First posted 2015-10-15 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Indolent Non-Hodgkin's Lymphoma; Follicular Lymphoma; Small Lymphocytic Lymphoma; Marginal Zone Lymphoma
Keywords: Phase 3; iNHL; Follicular Lymphoma; FL; PI3K; Small Lymphocytic Lymphoma; SLL; Marginal Zone Lymphoma; MZL
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — duvelisib; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duvelisib + Rituximab + Bendamustine (Experimental): Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules.
  Bendamustine is administered as an intravenous (IV) infusion and is supplied for injection in single-use vials at two strengths, 25 mg and 100 mg.
  Rituximab is administered as an IV infusion and is supplied in single-use vials at two strengths, 100 mg and 500 mg.
  Interventions: Drug: Duvelisib; Drug: Rituximab; Drug: Bendamustine
- Placebo + Rituximab + Bendamustine (Placebo Comparator): Placebo is administered orally and supplied as formulated capsules to match the active 5 mg and 25 mg capsules of duvelisib.
  Bendamustine is administered as an IV infusion and is supplied for injection in single-use vials at two strengths, 25 mg and 100 mg.
  Rituximab is administered as an IV infusion and is supplied in single-use vials at two strengths, 100 mg and 500 mg.
  Interventions: Drug: Placebo; Drug: Rituximab; Drug: Bendamustine

INTERVENTIONS:
Drug: Duvelisib — Duvelisib (25 mg BID) administered orally in 28-day continuous treatment cycles
  Other Names: IPI-145
  Arms: Duvelisib + Rituximab + Bendamustine
Drug: Placebo — Matching placebo (25 mg BID) administered orally in 28-day continuous treatment cycles
  Arms: Placebo + Rituximab + Bendamustine
Drug: Rituximab — IV infusion of rituximab (375 mg/m2) on Day 1 of Cycles 1-6.
  Other Names: Rituxan; MabThera
Drug: Bendamustine — IV infusion of bendamustine (90 mg/m2) on Day 1 and Day 2 of Cycles 1-6.
  Other Names: Treanda; Levact

SUMMARY:
This study will evaluate the efficacy and safety of duvelisib in combination with bendamustine and rituximab (DBR) vs placebo in combination with bendamustine and rituximab (PBR) in subjects with previously-treated indolent non-Hodgkin lymphoma (iNHL).

DETAILED DESCRIPTION:
Study IPI-145-22 is an international, multicenter, randomized, double-blind, placebo-controlled, two-arm Phase 3 study designed to evaluate efficacy and safety of DBR vs PBR in subjects with previously-treated iNHL (including follicular lymphoma [FL], small lymphocytic lymphoma [SLL] and marginal zone lymphoma [MZL]).

Approximately 600 subjects will receive 25 mg of duvelisib or placebo, orally BID for 28 day continuous cycles, in combination with 375 mg/m2 of rituximab given on Day 1 of Cycles 1-6 and 90 mg/m2 of bendamustine given on Day 1 and Day 2 of Cycles 1-6. Subjects will receive duvelisib until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of iNHL with one of the following histologic sub-types and grade:

  * Follicular lymphoma (FL)Grade 1, 2, or 3a
  * Small lymphocytic lymphoma (SLL)
  * Marginal zone lymphoma (MZL)( splenic, nodal, or extranodal)
* Have received the following systemic treatments for iNHL:

  * an anti-CD20 antibody; and
  * chemotherapy
* At least 1 measurable disease lesion > 1.5 cm in at least one dimension by computed tomography (CT)/CT-PET or magnetic resonance imaging (MRI)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2 (corresponds to Karnofsky Performance Status [(KPS) ≥60%])

Exclusion Criteria:

* Clinical evidence of transformation to a more aggressive subtype of lymphoma or grade 3B FL
* Refractory to bendamustine + rituximab therapy or single-agent bendamustine 120 mg/m2, with refractory defined as:

  - Progression of disease while receiving or within 6 months of completing treatment
* Severe allergic or anaphylactic reaction to any monoclonal antibody therapy, murine protein, or known hypersensitivity to any of the study drugs
* Received prior allogeneic transplant
* Received prior treatment with a phosphoinositide-3-kinase (PI3K) inhibitor
* Infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* History of tuberculosis treatment within the two years prior to randomization
* History of chronic liver disease, veno-occlusive disease, or alcohol abuse
* Ongoing treatment with chronic immunosuppressants (e.g., cyclosporine) or systemic steroids > 20 mg of prednisone (or equivalent) daily (QD)
* Ongoing treatment for systemic bacterial, fungal, or viral infection at screening
* Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), or herpes zoster (VZV) at screening
* Concurrent active malignancy other than adequately treated non-melanoma skin cancer or lentigo maligna without evidence of invasive disease or adequately treated cervical carcinoma in situ without evidence of disease
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or a pacemaker within the last 6 months prior to screening
* History of progressive multifocal leukoencephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From date of enrollment until the date of first documentation of progression or date of death from any cause, whatever came first, assessed up to 78 months

SECONDARY OUTCOMES:
Complete Response (CRR) | Every 3-6 Cycles (each cycle is 28 days) from date of randomization, until date of first documented progression. Subjects will be evaluated for progression through the primary analysis of the study or 5 years from randomization, whichever is later.
Overall Response Rate (ORR) | Every 3-6 Cycles (each cycle is 28 days) from date of randomization, until date of first documented progression. Subjects will be evaluated for progression through the primary analysis of the study or 5 years from randomization, whichever is later.
Overall Survival (OS) | Every 6 months for up to 5 years from date of randomization
Duration of Response (DOR) | Every 3-6 Cycles (each cycle is 28 days) from date of randomization, until date of first documented progression. Subjects will be evaluated for progression through the primary analysis of the study or 5 years from randomization, whichever is later.
Safety (Treatment- emergent adverse events (TEAEs) and changes in safety laboratory values) | Continuous from informed consent until 30 days from last dose
Pharmacokinetics (PK) | Cycle 1 and Cycle 2 (each cycle is 28 days)
  Evaluate the Duvelisib concentration in plasma sample.
Pharmacokinetics (PK) | Cycle 1 and Cycle 2 (each cycle is 28 days)
  Evaluate IPI-656 (metabolite) concentration in plasma sample.

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (7):
- United States (7):
  - Plainville, Connecticut
  - Plantation, Florida
  - Thomasville, Georgia
  - East Setauket, New York
  - Cookeville, Tennessee
  - Knoxville, Tennessee
  - Spokane, Washington